CLINICAL TRIAL: NCT02646566
Title: Randomised, Double-blind, Placebo-controlled Study of APD421 (Amisulpride for IV Injection) as Treatment of Established Post-operative Nausea and Vomiting, in Patients Who Have Had Prior Prophylaxis
Brief Title: Study of APD421 as PONV Treatment (Prior Prophylaxis)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DP10019
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- APD421 standard (Experimental): Single (standard) dose IV APD421
  Interventions: Drug: APD421
- APD421 high (Experimental): Single (high) dose IV APD421
  Interventions: Drug: APD421
- Placebo (Placebo Comparator): Single IV placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APD421
  Arms: APD421 high; APD421 standard
Drug: Placebo
  Arms: Placebo

SUMMARY:
Double-blind, randomised, parallel-group, placebo-controlled, adaptive, seamless, dose-selecting study to compare the efficacy of APD421 to placebo as treatment of established PONV, in patients who have had prior PONV prophylaxis.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients ≥ 18 years of age
* Provision of written informed consent
* Patients scheduled to undergo elective surgery (open or laparoscopic technique) under general anaesthesia (other than total intravenous anaesthesia with propofol) expected to last at least one hour from induction of anaesthesia to extubation
* Patients judged by the investigator to have a moderate or high risk of experiencing PONV. In forming this judgment, investigators should pay particular attention to risk factors such as a past history of PONV and/or motion sickness; habitual non-smoking status; female sex; and likely use of opioid analgesia post-operatively.
* For females of child-bearing potential: ability and willingness to use a highly effective form of contraception (as defined in ICH M3 guidance, e.g., abstinence from sexual intercourse, surgical sterilisation (of subject or partner), combined oral contraceptive pill, a double-barrier method of contraception such as either an intra-uterine device (IUD) or an occlusive cap with spermicide, in conjunction with partner's use of a condom, or any other method or combination of methods with a failure rate generally considered to be <1% per year) between the date of screening and at least 48 hours after administration of study drug
* In order to be eligible for randomisation, subjects must also:

  (i) have experienced a first episode of PONV not more than 24 hours after the end of their operation (wound closure) and prior to discharge from hospital ("qualifying PONV episode"), for which they have not already received any anti-emetic treatment; and (ii) not have received any dopamine-antagonist agent likely to prevent or treat nausea or vomiting (given as prophylaxis or otherwise) in the period from 24 hours prior to the start of their operation up to the time of the qualifying PONV episode.

Exclusion Criteria:

* Patients scheduled to undergo transplant surgery or any surgery where post-operative emesis may pose a significant danger to the patient
* Patients planned to receive only a local anaesthetic and/or regional neuraxial (intrathecal or epidural) block
* Patients who have received APD421 active ingredient for any indication within the last 2 weeks
* Patients who are allergic to APD421 active ingredient or any of the excipients of APD421
* Patients with a significant, ongoing history of vestibular disease or dizziness
* Patients with a known prolactin-dependent tumour (e.g. pituitary gland prolactinoma or breast cancer) or phaeochromocytoma.
* Patients with documented or suspected alcohol or substance abuse within the past 6 months.
* Patients with direct or indirect evidence of clinically significant hypokalaemia, such as a serum potassium level < 3.0 mmol/L.
* Patients who have received in the post-operative period, and prior to receiving study drug, any medication with a substantial risk of inducing torsades de pointes, including Class Ia antiarrhythmic agents such as quinidine, disopyramide, procainamide; Class III antiarrhythmic agents such as amiodarone and sotalol; and other medications such as bepridil, cisapride, thioridazine, methadone, IV erythromycin, IV vincamine, halofantrine, pentamidine, sparfloxacin, etc.
* Patients who have a documented, clinically significant cardiac arrhythmia or congenital long QT syndrome.
* Patients who are pregnant or breast feeding.
* Patients being treated with levodopa.
* Patients diagnosed with Parkinson's disease.
* Patients who have received emetogenic anti-cancer chemotherapy in the previous 4 weeks.
* Patients with a history of epilepsy.
* Any other concurrent disease or illness that, in the opinion of the investigator makes the patient unsuitable for the study.
* Patients who have previously participated in this study or who have participated in another interventional clinical study involving pharmacological therapy within the previous 28 days (or longer exclusion period, if required by national or local regulations).
* Where local laws/regulations require: patients under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Fox, MB BChir, Study Director — Acacia Pharma Ltd
Locations (8):
- United States (4):
  - Jackson Memorial Hospital, Miami, Florida
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
- CHU de Hautepierre, Strasbourg, France
- Germany (3):
  - HELIOS Klinikum Aue, Aue
  - Universität Heidelberg, Heidelberg
  - Philipps University, Marburg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Estimated recruitment was 700, to deliver 690 evaluable, randomised patients, providing an average of 230 evaluable patients in each of the three groups. The number of randomised patients planned per country was as follows: Germany, 190; France, 15; Canada, 100; and USA, 395
Pre-assignment Details: Three patients were randomised but not dosed: 2 due to withdrawal of consent, 1 for other reasons.
Groups:
- APD421 5mg: APD421 5mg administered as a single, slow intravenous (IV) push over about two minutes
- APD421 10mg: APD421 10mg administered as a single,slow intravenous (IV) push over about two minutes
- Placebo: Matching Placebo administered as a single, slow intravenous (IV) push over about two minutes
Period: Overall Study
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Started | 237 | 230 | 235
Completed | 231 | 226 | 230
Not Completed | 6 | 4 | 5
Not completed — Lost to Follow-up | 5 | 4 | 5
Not completed — Treatment failure | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- APD421 10mg: APD421 10mg administered as a single, slow intravenous (IV) push over about two minutes
- Placebo: Matching placebo administered as a single, slow, IV push over about two minutes
- Total: Total of all reporting groups
Arm/Group | APD421 5mg | APD421 10mg | Placebo | Total
Number analyzed (Participants) | 237 | 230 | 235 | 702
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 1 | 4
  Between 18 and 65 years | 214 | 204 | 216 | 634
  >=65 years | 22 | 24 | 18 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.8 (13.12) | 46.9 (13.03) | 46.0 (13.38) | 46.3 (13.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213 | 208 | 212 | 633
  Male | 24 | 22 | 23 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 5 | 6 | 8 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 19 | 21 | 22 | 62
  White | 196 | 189 | 193 | 578
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 15 | 14 | 12 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response (Success of Initial PONV Treatment)
Description: The primary efficacy variable was the dichotomous variable: success or failure of initial PONV treatment, where success is defined as no emetic episodes (vomiting or retching) from 30 minutes* to 24 hours after administration of study medication and no administration of anti-emetic rescue medication at any time in the 24-hour period after administration of study medication.
Time Frame: 0-24 hours after administration of study medication
Population: Modified ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 237 | 230 | 235
Participants | 80 | 96 | 67
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; The primary efficacy analysis was a comparison of the incidence of the primary efficacy variable between the two groups that received APD421 and the group that received placebo, using Pearson's χ2 test. The threshold for determining statistical significance in the comparison of incidence of success between the active and placebo groups (the primary efficacy analysis) was a p-value of 2.5% one-sided; Test type: Superiority; p = 0.003, Chi-squared — One-sided p-value. After adjustment for multiplicity using Hommel's method. (Note: unadjusted p value = 0.003) A priori threshold for statistical significance = 0.025
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.109, Chi-squared — One-sided p-value. After adjustment for multiplicity using Hommel's method. (Note: unadjusted p value = 0.109) A priori threshold for statistical significance = 0.025

2. Secondary Outcome: Number of Participants With Complete Response 0-2 Hrs
Description: Success of initial PONV treatment, where success is defined as no emetic episodes (vomiting or retching) from 30 minutes* to 2 hours after administration of study medication and no administration of anti-emetic rescue medication at any time in the 2-hour period after administration of study medication.
Time Frame: 0-2 hours after administration of study medication
Population: Modified ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 237 | 230 | 235
Participants | 134 | 160 | 116
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p < 0.001, Chi-squared — One-sided p-value. No adjustment for multiple comparisons. A priori threshold for statistical significance = 0.025
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.059, Chi-squared — One-sided p-value. No adjustment for multiple comparisons. A priori threshold for statistical significance = 0.025

3. Secondary Outcome: Number of Participants With Complete Response 0-4 Hrs
Description: Success of initial PONV treatment, where success is defined as no emetic episodes (vomiting or retching) from 30 minutes* to 4 hours after administration of study medication and no administration of anti-emetic rescue medication at any time in the 4-hour period after administration of study medication.
Time Frame: 0-4 hours after administration of study medication
Population: Modified ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 237 | 230 | 235
Participants | 105 | 136 | 87
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p < 0.001, Chi-squared — One-sided p-value. No adjustment for multiple comparisons. A priori threshold for statistical significance = 0.025
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.053, Chi-squared — One-sided p-value. No adjustment for multiple comparisons. A priori threshold for statistical significance = 0.025

4. Secondary Outcome: Number of Participants With Complete Response 0-6 Hrs
Description: Success of initial PONV treatment, where success is defined as no emetic episodes (vomiting or retching) from 30 minutes to 6 hours after administration of study medication and no administration of anti-emetic rescue medication at any time in the 6-hour period after administration of study medication.
Time Frame: 0-6 hours after administration of study medication
Population: Modified ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 237 | 230 | 235
Participants | 99 | 121 | 77
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p < 0.001, Chi-squared — One-sided p-value. No adjustment for multiple comparisons. A priori threshold for statistical significance = 0.025
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.021, Chi-squared — One-sided p-value. No adjustment for multiple comparisons. A priori threshold for statistical significance = 0.025

5. Secondary Outcome: Time to Treatment Failure
Description: Time to first violation of the criteria for complete response
Time Frame: 0-24 hours after study drug administration
Population: Modified ITT population
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 237 | 230 | 235
minutes | 188 [43 to NA] — Treatment failure occurred in less than 75% of patients | 443 [70 to NA] — Treatment failure occurred in less than 75% of patients | 120 [35 to NA] — Treatment failure occurred in less than 75% of patients
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Cox
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.084, Regression, Cox

6. Secondary Outcome: Number of Patients With Incidence of Emesis
Description: Number of patients experiencing vomiting or retching during the time period from 30 minutes to 24 hours after administration of study medication
Time Frame: 30 mins to 24 hours after study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 237 | 230 | 235
Participants | 43 | 36 | 67
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.004, Chi-squared

7. Secondary Outcome: Number of Patients Receiving Rescue Medication
Description: Number of patients receiving pre-specified anti-emetic rescue medication at any time in the 24 hours post-treatment period
Time Frame: 0-24 hours after study drug administration
Population: Modified ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 237 | 230 | 235
Participants | 155 | 127 | 163
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.179, Chi-squared

8. Secondary Outcome: Number of Patients With an Incidence of Significant Nausea
Description: Number of patients with nausea score ≥4 on an 11-point verbal rating scale (0=no nausea, 10=worst possible nausea, therefore higher value is worse outcome) during the time period from 30 minutes to 24 hours after administration of study medication.
Time Frame: 30 mins to 24 hours after study drug administration
Population: Modified ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 237 | 230 | 235
Participants | 135 | 111 | 139
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p = 0.009, Chi-squared
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.315, Chi-squared

9. Secondary Outcome: Number of Patients With an Incidence of Nausea
Description: Number of patients with nausea score ≥1 on an 11-point verbal rating scale (0=no nausea, 10=worst possible nausea, therefore higher value is worse outcome) during the time period from 30 minutes to 24 hours after administration of study medication.
Time Frame: 30 mins to 24 hours after drug administration
Population: Modified ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 237 | 230 | 235
Participants | 183 | 163 | 181
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p = 0.065, Chi-squared
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.520, Chi-squared

10. Secondary Outcome: Maximum Severity of Nausea
Description: Highest recorded nausea score on an 11-point verbal rating scale (0=no nausea, 10=worst possible nausea, therefore higher value is worse outcome) during the time period from 30 minutes to 24 hours after administration of study medication.
Time Frame: 30 mins to 24 hours after study drug administration
Population: Modified ITT population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 237 | 230 | 235
Score on a scale | 4.1 (3.08) | 3.6 (3.03) | 4.2 (3.04)
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.420, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Evolution Score of Nausea (0-180 Mins)
Description: The evolution score of nausea was calculated as the area under the curve (AUC) of the nausea scores on a scale 0-10 (where 0 is no nausea and 10 is the worst nausea imaginable) obtained at five pre-planned time points: pre-dose (0-min), and 5, 15 and 30 minutes and 2 hours after administration of study medication, as well as any spontaneously reported episodes of nausea during the time period, plotted against time. A higher score represents a worse outcome.
Time Frame: 0-180 minutes after study drug administration
Population: Modified ITT population
Measure: Mean (Standard Deviation); unit: Score on a scale*min
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 237 | 230 | 235
Score on a scale*min | 6994.7 (5659.6) | 5637.9 (6046.6) | 7629.2 (6640.2)
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.258, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 7 days
Description: Any AE that is serious, occurring during the relevant study period (from study drug administration to 7-day follow-up), irrespective of the treatment received by the subject, must be reported to the Pharmacovigilance provider within 24 hours
Groups:
- APD421 IV 5mg: IV dose of APD421 5mg (IV dose)- was administered to each patient in a double-blind fashion, by slow IV push over about two minutes into a peripheral or central venous cannula.
- APD421 IV 10mg: IV dose of APD421 10mg (IV dose)- was administered to each patient in a double-blind fashion by slow IV push over about two minutes into a peripheral or central venous cannula.
- Placebo: IV dose of Placebo (IV dose)- was administered to each patient in a double-blind fashion by slow IV push over about two minutes into a peripheral or central venous cannula.
Arm/Group | APD421 IV 5mg | APD421 IV 10mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/237 | 0/230 | 0/235
Serious Adverse Events (participants affected / at risk) | 6/237 | 3/230 | 5/235
Other Adverse Events (participants affected / at risk) | 64/237 | 66/230 | 78/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APD421 IV 5mg (N=237) | APD421 IV 10mg (N=230) | Placebo (N=235)
Anastomosis Insufficiency (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Non-infectious gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Unspecified Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal Hematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intractable vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Abscess Presacral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fatty tissue prolapse at the tempral lobe (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Numbness in the leg (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Postoperative rise in creatinine (Investigations) | 1 (1) | 0 (0) | 0 (0)
Post cholecystectomy bile leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Postoperative Ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APD421 IV 5mg (N=237) | APD421 IV 10mg (N=230) | Placebo (N=235)
Nausea (Gastrointestinal disorders) | 30 (33) | 27 (28) | 30 (32)
Flatulence (Gastrointestinal disorders) | 13 (13) | 13 (13) | 18 (18)
Constipation (Gastrointestinal disorders) | 13 (13) | 11 (11) | 17 (17)
Vomiting (Gastrointestinal disorders) | 11 (14) | 10 (11) | 13 (13)
Headache (Nervous system disorders) | 10 (10) | 10 (10) | 17 (17)
Infusion site pain (General disorders) | 8 (8) | 12 (12) | 10 (10)
Pruritus (General disorders) | 7 (7) | 10 (10) | 13 (13)

LIMITATIONS AND CAVEATS:
There were no limitations or caveats with this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No